CLINICAL TRIAL: NCT06823154
Title: The Implementation and Impact of an Allergy De-Labeling Program in the Emergency Department: The De-Label Program Expansion
Brief Title: The Implementation and Impact of an Allergy De-Labeling Program in the Emergency Department
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Staff physician, Principal Investigator, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000069700
Record Dates: First submitted 2024-06-25; First posted 2025-02-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Allergy Amoxicillin; Beta-lactam Allergy Labels
Keywords: Beta-lactam allergy labels; Pediatrics; Oral challenge; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eligible for study risk assessment questionnaire (Experimental): First, a systematic allergy risk assessment tool will enable stratification of patients' reported symptoms as (1) low risk (eg, isolated urticarial, maculopapular rash, gastrointestinal symptoms) or (2) high risk (eg, anaphylaxis, severe systemic reactions). Only patients classified low risk will be eligible for OPC for allergy delabeling. Patients' ineligible for OPC because of history of high-risk allergy symptoms or presence of clinical confounders for OPC (eg, uncontrolled asthma) will be referred to the SickKids allergy clinic for further evaluation.
  Interventions: Other: Study questionnaire
- Eligible for oral challenge in the emergency department (Experimental): A subset of patients screened with the risk assessment questionnaire will fulfill eligibility criteria to undergo the Oral provocation challenge. Specifically, these will be patients who (1) fulfill several procedural requirements (eg, parent able to observe child for 1 hour after OPC), (2) have a previously unevaluated allergy label without high-risk features and without any clinical confounders for the OPC, and (3) meet other clinical criteria for OPC (eg, vital signs within normal range). These participants will be given a one-time dose of Amoxicillin 17 mg/kg (maximum, 500 mg) and observed for 1 hour for a reaction.
  Interventions: Drug: Amoxicillin; Other: Study questionnaire

INTERVENTIONS:
Drug: Amoxicillin — Prospective cohort study of patients presenting to the ED with a reported BLA. (1) Allergy history and risk assessment, (2) Oral provocation challenge (if eligible), and (3) Post-discharge follow-up (if received OPC or referred to allergy).
  Arms: Eligible for oral challenge in the emergency department
Other: Study questionnaire — In the first component of the study, research staff will survey patients for history pertinent to their BLA label. This includes questions regarding any prior evaluations, patients' perception of their allergy label, and clinical details of allergy history. The latter involves an allergy history risk assessment, which will screen patient for high-risk features (eg, new maculopapular rash within 2 hours of administering antibiotic). Presence of any high-risk features will disqualify the patient from subsequent study components.
  Finally, the questionnaire will screen for presence of any clinical confounders that would preclude administration of the OPC (eg, use of antihistamines within prior 72 hours).

SUMMARY:
Beta-lactams are the most common antibiotics prescribed to children, including penicillin and amoxicillin. They are usually more effective and have fewer side effects than other ty antibiotics. Some children can have reactions to these antibiotics that can be mistaken as an allergy, especially rashes that develop days to weeks later. In such cases, when children take the antibiotic again, they have no problem tolerating it; this is called "delabeling an allergy" with an "oral challenge". Based on our experience with a similar program among inpatients, we are implementing and evaluating an allergy delabeling program for children in the SickKids ED, with the hope and intent to delabel most children of their "allergies" using an oral challenge.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients aged 1 month to 18 years who present to the SickKids ED with a reported BLA will be eligible for the allergy history component of the study.

Exclusion Criteria:

* Parent/guardian and/or patient unable to consent or assent.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the proportion of patients delabeled among those given the OPC. | Up to 2 weeks
  In the primary analysis, successful BLA removal will be defined as tolerating OPC without any immediate adverse reaction.

SECONDARY OUTCOMES:
The proportion of patients with a reported BLA who are low risk (potential impact) | Day 1
  This includes questions regarding any prior evaluations, patients' perception of their allergy label, and clinical details of allergy history. The latter involves an allergy history risk assessment, which will screen patient for high-risk features (eg, new maculopapular rash within 2 hours of administering antibiotic). Presence of any high-risk features will disqualify the patient from subsequent study components.
  Finally, the questionnaire will screen for presence of any clinical confounders that would preclude administration of the OPC (eg, use of antihistamines within prior 72 hours).
The proportion of patients successfully delabeled without any adverse reactions (immediate or delayed up to 2 weeks) | Up to 2 weeks
  Successful BLA removal will be defined as tolerating OPC without any immediate adverse reaction.
The proportion of patients who receive or are prescribed amoxicillin or a first-generation cephalosporin, among patients who undergo OPC | Day 1
Feasibility based on proportion of eligible participants who consent to OPC | Up to 2 weeks
Feasibility based on duration of allergy risk assessment and OPC (calculated using CRF timestamps) | Up to 2 weeks
Patient and caregiver perspectives on BLA and OPC | Day 1
  After completion of the oral challenge, participants and their caregivers will complete a study questionnaire to assess their opinions about the safety of the oral challenge and their comfortability with having the allergy label removed from their chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Monica Caldeira-Kulbakas, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No